CLINICAL TRIAL: NCT00932737
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group Pilot Study of the Efficacy and Safety of Oral Doses of 20 mg Hyoscine Butylbromide When Used on Demand for the Treatment of Self-reported Functional Abdominal Pain Associated With Cramping
Brief Title: (Hyoscine Butylbromide) for Abdominal Pain Associated With Cramping on Demand Basis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202.839; U09-3181-01
Record Dates: First submitted 2009-06-17; First posted 2009-07-03 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — beta-Globins

ARMS (2):
- Hyoscine butylbromide (HBB) 20mg 1-5 tablets per episode (Active Comparator): Patient to receive 1-5 tablets containing 20mg HBB per Abdominal pain associated with cramping (APC) episode
  Interventions: Drug: HBB 20 mg
- Placebo (Placebo Comparator): patient to receive a tablet identical to those containing HBB and take 1-5 tablets per episode
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 1-5 tablets per episode
  Arms: Placebo
Drug: HBB 20 mg — Active drug, one to five tablets per episode
  Arms: Hyoscine butylbromide (HBB) 20mg 1-5 tablets per episode

SUMMARY:
The primary objective of this pilot study is to assess effects of Hyoscine Butylbromide (HBB) 20 mg in comparison to placebo, when used as needed, as measured by the subject's assessment of intensity of abdominal pain associated with cramping (APC) in the treatment of two episodes.

ELIGIBILITY:
Inclusion Criteria:

History of recurrent abdominal pain with cramping (APC) for at least three months.

Recorded at least two episodes of APC of at least "moderate" intensity (i.e., 5 or above on a 0-10 point scale) lasting one hour in the eDiary during the run-in period.

Exclusion Criteria:

Experiencing daily episode of APC during Run-in period Active gastrointestinal disease during the past 12 months including malignancy, inflammatory bowel disease, celiac disease or complete or partial bowel obstruction and who have undergone major gastrointestinal surgery with the past 12 months (patients with history of appendectomy, cholecystectomy, bilateral tubal ligation and c-section within past 12 months are allowed in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2009-06-09 (Actual); Primary Completion 2010-02-08 (Actual); Study Completion 2010-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (19):
  - 202.839.01014 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 202.839.01003 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 202.839.01001 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 202.839.01002 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 202.839.01017 Boehringer Ingelheim Investigational Site, Rockford, Illinois
  - 202.839.01005 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 202.839.01019 Boehringer Ingelheim Investigational Site, Chevy Chase, Maryland
  - 202.839.01009 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 202.839.01004 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 202.839.01011 Boehringer Ingelheim Investigational Site, Toms River, New Jersey
  - 202.839.01008 Boehringer Ingelheim Investigational Site, Lake Success, New York
  - 202.839.01015 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 202.839.01021 Boehringer Ingelheim Investigational Site, Norman, Oklahoma
  - 202.839.01010 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 202.839.01013 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 202.839.01006 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 202.839.01012 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 202.839.01007 Boehringer Ingelheim Investigational Site, Virginia Beach, Virginia
  - 202.839.01020 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, placebo-controlled, randomized, parallel-group pilot study aimed to assess the efficacy and safety of oral doses of 20 milligram hyoscine butylbromide when used on demand for the treatment of abdominal pain associated with cramping over a treatment period of 4 weeks.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. 22 enrolled subjects didn't receive any trial medication
Groups:
- Placebo: Up to 5 film-coated tablets of 20 milligram (mg) matching placebo (Tota up to 100 mg) were administered orally per episode. One or two episodes of Abdominal pain associated with cramping (APC) were treated up to 2 hours each within 4 weeks.
- Hyoscine Butylbromide (Buscopan®) 20 mg: Up to 5 film-coated tablets of 20 milligram (mg) of Hyoscine butylbromide (Buscopan®) (Total up to 100 mg) were administered orally per episode. One or two episodes of Abdominal pain associated with cramping (APC) were treated up to 2 hours each within 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Started | 87 | 88
Completed | 86 | 87
Not Completed | 1 | 1
Not completed — Not treated in second episode | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: This patient set includes all randomized patients who were dispensed study medication during treatment period and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (11.3) | 39.7 (15.0) | 38.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 130
  Male | 19 | 26 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 34 | 67
  White | 52 | 54 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Numeric pain rating scale (NPRS) for intensity of APC in episode 1 [Mean (Standard Deviation); unit: Score on a scale] — The intensity of Abdominal pain associated with cramping (APC) was rated on an 11-point numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
  Score on a scale | 7.67 (1.67) | 7.57 (1.42) | 7.62 (1.55)
Numeric pain rating scale (NPRS) for intensity of APC in episode 2 [Mean (Standard Deviation); unit: Score on a scale] — The intensity of Abdominal pain associated with cramping (APC) was rated on an 11-point numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Population: Full analysis set (FAS): This patient set includes all treated patients who experienced at least one episode of Abdominal pain associated with cramping (APC) and took at least one dose of study medication to treat the symptoms and had baseline rating of APC in that episode over a four week period following randomization. Participants with non-missing values were included.
  Score on a scale
    number analyzed (Participants) | 72 | 78 | 150
    (all) | 7.86 (1.51) | 7.73 (1.44) | 7.79 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intensity of Abdominal Pain Associated With Cramping Following Treatment Based on the Numeric Pain Rating Scale (NPRS) in Episode 1
Description: The intensity of Abdominal pain associated with cramping was rated on an 11-point numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: At baseline (prior to intake of first tablet of study medication in episode 1) until 4 hours thereafter or until the patient had responded that their pain was absent, up to 4 hours
Population: Full analysis set (FAS): This patient set includes all treated patients who experienced at least one episode of Abdominal pain associated with cramping (APC) and took at least one dose of study medication to treat the symptoms and had baseline rating of APC in that episode over a four week period following randomization.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Score on a scale | -2.7 (3.10) | -3.1 (3.05)
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; A model included fixed, categorical effects of treatment group, episode, interval and center, as well as the treatment-by-episode interaction, with the covariate of baseline intensity of Abdominal pain associated with cramping . An unstructured covariance structure was used to model the within-patient errors; Test type: Other; p = 0.0156, Mixed effect model; Adjusted mean difference = -0.7, 95% CI 2-sided [-1.3 to -0.1], Standard Error of Mean 0.29 — The adjusted mean difference between Hyoscine butylbromide minus Placebo was calculated

2. Primary Outcome: Change From Baseline in Intensity of Abdominal Pain Associated With Cramping Following Treatment Based on the Numeric Pain Rating Scale (NPRS) in Episode 2
Description: as for outcome 1
Time Frame: At baseline (prior to intake of first tablet of study medication in episode 2) until 4 hours thereafter or until the patient had responded that their pain was absent, up to 4 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 72 | 78
Score on a scale | -2.9 (3.15) | -3.2 (3.06)
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0512, Mixed effect model; Adjusted mean difference = -0.6, 95% CI 2-sided [-1.2 to 0.0], Standard Error of Mean 0.30 — The adjusted mean difference between Hyoscine butylbromide minus Placebo was calculated

3. Primary Outcome: Area Under the Curve (AUC) Calculated From the Responses to the Numeric Pain Rating Scale (NPRS) Scores in Episode 1
Description: as for outcome 1
Time Frame: At baseline (prior to intake of first tablet of study medication for episode 1) and 15 minutes(min), 30min, 45min, 1 hour(h), 1h30min, 2h, 2h30min, 3h, 3h30min, and 4h thereafter.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score * hours
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Score * hours | -3.71 (2.42) | -4.32 (2.27)
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; The analysis of covariance (ANCOVA) was performed on the change from baseline to the last recorded rating of intensity for each treated episode of Abdominal pain associated with cramping (APC). The statistical model included the main effects of treatment, episode, and center as well as terms for the treatment-by-episode interaction, with baseline intensity of APC for the respective episode as a covariate; Test type: Other; p = 0.0351, ANCOVA; Adjusted mean difference = -0.7, 95% CI 2-sided [-1.3 to 0.0], Standard Error of Mean 0.32 — The adjusted mean difference between Hyoscine butylbromide minus Placebo was calculated

4. Primary Outcome: Area Under the Curve (AUC) Calculated From the Responses to the Numeric Pain Rating Scale (NPRS) Scores in Episode 2
Description: as for outcome 1
Time Frame: At baseline (prior to intake of first tablet of study medication for episode 2) and 15 minutes(min), 30min, 45min, 1 hour(h), 1h30min, 2h, 2h30min, 3h, 3h30min, and 4h thereafter.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score * hours
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 72 | 78
Score * hours | -4.17 (2.51) | -4.40 (2.32)
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.3557, ANCOVA; Adjusted mean difference = -0.3, 95% CI 2-sided [-1.0 to 0.4], Standard Error of Mean 0.35 — The adjusted mean difference between Hyoscine butylbromide and Placebo was calculated

5. Primary Outcome: Percentage of Participants With Response of "no Pain" Based on Numeric Pain Rating Scale (NPRS) in Episode 1
Description: The intensity of Abdominal pain associated with cramping was rated on an 11-point numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Responses of "no pain" (NPRS = 0) based on the 0 to 10 point NPRS scale were summarized.
Time Frame: At 4 hours after intake of first tablet of study medication in episode 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Percentage of participants | 65.52 | 67.05
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.831, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 1.071, 95% CI 2-sided [0.572 to 2.004]

6. Primary Outcome: Percentage of Participants With Response of no Pain Based on Numeric Pain Rating Scale (NPRS) in Episode 2
Description: as for outcome 5
Time Frame: At 4 hours after intake of first tablet of study medication in episode 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 72 | 78
Percentage of participants | 69.44 | 71.79
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.557, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 1.222, 95% CI 2-sided [0.626 to 2.387]

7. Primary Outcome: Percentage of Participants With Response Based on the Patient Global Impression of Change (PGI-C) of "Much Better" in Episode 1
Description: At episode 1, after the intake of first tablet of study medication, the patient then responded to the question of "Compared to just before you took the first tablet of study medication, how would you rate your abdominal pain associated with cramping now?" based on the Patient global impression of change (PGI-C), using the available responses: "Much better", "Somewhat better", "A little better", "No change", "A little worse", and "Somewhat worse".
Time Frame: At 4 hours after intake of first tablet of study medication in episode 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Percentage of participants | 79.31 | 73.86
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.396, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 0.737, 95% CI 2-sided [0.365 to 1.490]

8. Primary Outcome: Percentage of Participants With Response Based on the Patient Global Impression of Change (PGI-C) of "Much Better" in Episode 2
Description: At episode 2, after the intake of first tablet of study medication, the patient then responded to the question of "Compared to just before you took the first tablet of study medication, how would you rate your abdominal pain associated with cramping now?" based on the Patient global impression of change (PGI-C), using the available responses: "Much better", "Somewhat better", "A little better", "No change", "A little worse", and "Somewhat worse".
Time Frame: At 4 hours after intake of first tablet of study medication in episode 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 72 | 78
Percentage of participants | 76.39 | 80.77
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.448, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 1.336, 95% CI 2-sided [0.632 to 2.827]

9. Primary Outcome: Percentage of Participants With Response Based on the 4-point Verbal Rating Scale (VRS) of "Very Satisfied" in Episode 1
Description: At episode 1, after the intake of first tablet of study medication, the patient then responded to the question of "Overall, how satisfied were you with the medication in terms of effectiveness for this episode?" based on the 4-point Verbal rating scale (VRS) using the available response: "Very Satisfied", "Satisfied", "Dissatisfied", and "Very Dissatisfied".
Time Frame: At 4 hours after intake of first tablet of study medication in episode 1
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 76 | 69
Percentage of participants | 15.79 | 30.43
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.030, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 2.474, 95% CI 2-sided [1.093 to 5.604]

10. Primary Outcome: Percentage of Participants With Response Based on the 4-point Verbal Rating Scale (VRS) of "Very Satisfied" in Episode 2
Description: At episode 2, after the intake of first tablet of study medication, the patient then responded to the question of "Overall, how satisfied were you with the medication in terms of effectiveness for this episode?" based on the 4-point Verbal rating scale (VRS) using the available response: "Very Satisfied", "Satisfied", "Dissatisfied", and "Very Dissatisfied".
Time Frame: At 4 hours after intake of first tablet of study medication in episode 2
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 65 | 60
Percentage of participants | 32.31 | 43.33
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.167, Regression, Logistic; Logistic regression included the main effects of treatment group, episode, and center; Odds Ratio (OR) = 1.654, 95% CI 2-sided [0.810 to 3.378]

11. Primary Outcome: Time to Relief in Episode 1
Description: Time from intake of first tablet of study medication to first response of "no pain" (numeric pain rating scale (NPRS) = 0) in episode 1.
Time Frame: From intake of first tablet of study medication up to 4 hours thereafter in episode 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Minutes | 172.0 [122.0 to 202.0] | 130.0 [120.0 to 150.0]
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.2560, Log Rank; Log rank test was used for comparison of Hyoscine butylbromide (Buscopan®) 20 mg group versus Placebo group

12. Primary Outcome: Time to Relief in Episode 2
Description: Time from intake of first tablet of study medication to first response of "no pain" (numeric pain rating scale (NPRS) = 0) in episode 2.
Time Frame: From intake of first tablet of study medication up to 4 hours thereafter in episode 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 72 | 78
Minutes | 150.0 [120.0 to 182.0] | 120.0 [107.0 to 158.0]
Statistical Analysis 1: Comparison: Placebo vs Hyoscine Butylbromide (Buscopan®) 20 mg; Test type: Other; p = 0.5179, Log Rank; Log rank test was used for comparison of Hyoscine butylbromide (Buscopan®) 20 mg group versus Placebo group

13. Primary Outcome: Number of Tablets of Study Medication Taken
Description: Number of tablets of study medication taken in each of the two episode.
Time Frame: From intake of first tablet of study medication up to 4 hours thereafter in each episode.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tablets
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Tablets
  Episode 1 | 3.5 (1.2) | 3.3 (1.3)
  Episode 2 | 3.1 (1.5) | 3.0 (1.4)

14. Secondary Outcome: Percentage of Patients With Drug-related Adverse Events
Time Frame: From the first dose of study medication until 3 days after the last dose for each episode. Up to 8 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
Percentage of participants | 4.6 | 3.4

15. Secondary Outcome: Number of Participants Per Verbal Rating Scale Assessing Participant's Global Assessment of Tolerability in Episode 1
Description: Patient's global assessment of tolerability following treatment of an episode of Abdominal pain associated with cramping (APC) was based on a 4-point Verbal rating scale (VRS) in patient's response to the question, "Overall, how satisfied were you with the medication in terms of side effects during this episode?" ("Very Satisfied," "Satisfied," "Dissatisfied," "Very Dissatisfied").
Time Frame: At 4 hours after intake of first tablet of study medication in episode 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 76 | 69
Participants
  Very satisfied | 24 | 36
  Satisfied | 45 | 29
  Dissatisfied | 7 | 4
  Very dissatisfied | 0 | 0

16. Secondary Outcome: Number of Participants Per Verbal Rating Scale Assessing Participant's Global Assessment of Tolerability in Episode 2
Description: as for outcome 15
Time Frame: At 4 hours after intake of first tablet of study medication in episode 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 65 | 60
Participants
  Very satisfied | 27 | 34
  Satisfied | 34 | 25
  Dissatisfied | 3 | 1
  Very dissatisfied | 1 | 0

17. Secondary Outcome: Change From Baseline to End of Study Visit in Systolic Blood Pressure
Description: Change from baseline (intake of the first tablet of trial medication in the study) to end of study visit in systolic blood pressure.
Time Frame: At baseline (intake of the first tablet of trial medication in the study) and day 28 (end of study visit)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
millimetre of mercury (mmHg) | 2.52 (11.79) | -0.76 (10.84)

18. Secondary Outcome: Change From Baseline to End of Study Visit in Diastolic Blood Pressure
Description: Change from baseline (intake of the first tablet of trial medication in the study) to end of study visit in diastolic blood pressure.
Time Frame: At baseline (intake of the first tablet of trial medication in the study) and day 28 of end of study visit
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
millimetre of mercury (mmHg) | 0.21 (7.19) | 0.82 (8.37)

19. Secondary Outcome: Change From Baseline to End of Study Visit in Pulse Rate
Description: Change from baseline (intake of the first tablet of trial medication in the study) to end of study visit in pulse rate.
Time Frame: At baseline (intake of the first tablet of trial medication in the study) and day 28 of end of study visit
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
beats per minute (bpm) | -0.9 (11.1) | 0.8 (9.1)

20. Secondary Outcome: Change From Baseline to End of Study Visit in Body Temperature
Description: Change from baseline (intake of the first tablet of trial medication in the study) to end of study visit in body temperature.
Time Frame: At baseline (intake of the first tablet of trial medication in the study) and day 28 of end of study visit
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
celsius | -0.053 (0.508) | -0.036 (0.367)

21. Secondary Outcome: Change From Baseline to End of Study Visit in Respiratory Rate
Description: Change from baseline (intake of the first tablet of trial medication in the study) to end of study visit in respiratory rate.
Time Frame: At baseline (intake of the first tablet of trial medication in the study) and day 28 of end of study visit
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
Number analyzed (Participants) | 87 | 88
breaths per minute | 0.0 (2.4) | 0.2 (2.2)

ADVERSE EVENTS:
Time Frame: From first dose until end of study visit + 3 days, up to 31 days for all-cause mortality; From first dose until 3 days after last dose for each episode, up to 8 days for (serious) adverse events.
Description: Treated set: This patient set included all randomized patients who were dispensed study medication during the treatment period and were documented to have taken at least one dose of investigational treatment. Any newly emergent abnormalities noted during the physical examination at the end of the study were recorded as adverse events and were reported together with adverse events.
Arm/Group | Placebo | Hyoscine Butylbromide (Buscopan®) 20 mg
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/87 | 1/88
Other Adverse Events (participants affected / at risk) | 0/87 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Hyoscine Butylbromide (Buscopan®) 20 mg (N=88)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.